CLINICAL TRIAL: NCT06746376
Title: Effect of a Specific Hand Intervention Program With Strength and Manipulative Dexterity Exercises in Women With Arthralgia Secondary to Hormone Therapy Following Breast Cancer.
Brief Title: Effect of a Specific Hand Intervention in Women With Arthralgia Secondary to Hormone Therapy Following Breast Cancer.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Vanesa Abuín, Asistant Professor, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HANDPROJECT001
Record Dates: First submitted 2024-12-17; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Arthralgia
MeSH Terms: conditions — Arthralgia | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluator will be blinded to the patient's allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Description:
  Participants assigned to the intervention group will undergo a 8-week supervised hand exercise program designed to improve pain, manual dexterity, and functionality. Sessions will last 45 minutes and occur once per week under the supervision of a qualified occupational therapist and one self-administrated home exercise session. The program includes three structured phases per session
  Warm-Up Phase (10 minutes)
  Gentle hand and wrist stretches Main Exercise Phase (25 minutes)
  This phase focuses on strengthening, manual dexterity, and functional tasks:
  Strengthening Exercises
  Manual Dexterity Exercises
  Functional Tasks (Simulated Activities of Daily Living - AVDs):
  Cool-Down Phase (10 minutes)
  8 weeks, with 45-minute sessions twice weekly.
  Interventions: Other: Occupational Therapy
- Control (No Intervention): Description:
  Participants in the control group will not receive any intervention during the study period. They will undergo the same assessments as the intervention group at baseline and after 8 weeks to evaluate changes over time.
  Details:
  The control group will serve as a comparison to determine the effects of time alone on pain, manual dexterity, and hand functionality in women with hormone therapy-related arthralgia.
  Participants will continue their usual daily activities and standard care during the study period.
  No specific exercises or additional therapies will be provided as part of the study.

INTERVENTIONS:
Other: Occupational Therapy — Description:
  Participants assigned to the intervention group will undergo a 8-week supervised hand exercise program designed to improve pain, manual dexterity, and functionality.
  Arms: Intervention

SUMMARY:
This study aims to evaluate the impact of a 12-week hand exercise program on pain, manual dexterity, and hand function in women experiencing hand joint pain (arthralgia) due to hormone therapy after breast cancer. Participants will be randomly assigned to either an intervention group, where they will perform specific hand exercises, or a control group, which will not receive any exercise program. Pain levels, hand function, and manual dexterity will be assessed before and after the intervention using questionnaires and functional tests. The goal is to determine whether targeted hand exercises can improve pain and daily hand use in this population.

DETAILED DESCRIPTION:
This is a randomized, evaluator-blinded clinical trial that aims to determine the effects of a 12-week hand exercise program on pain, manual dexterity, and functional performance in women experiencing hand arthralgia due to hormone therapy following breast cancer. Participants will be randomly assigned to one of two groups: an intervention group performing specific hand exercises or a control group with no exercise intervention.

The primary outcome will be changes in hand pain levels assessed using the Brief Pain Inventory (BPI) and McCaffrey's Initial Pain Assessment Tool. Secondary outcomes will include functional performance measured with the DASH and ABILHAND questionnaires, as well as manual dexterity, speed, and coordination assessed through standardized tests (Purdue Pegboard Test, Box and Block Test, and Minnesota Rate of Manipulation Test).

The study will evaluate the potential benefits of targeted hand exercises for improving pain, dexterity, and quality of life in breast cancer survivors experiencing treatment-related hand symptoms.

Detailed Description

Study Design:

Type: Interventional (Clinical Trial) Allocation: Randomized Intervention Model: Parallel Assignment Masking: Single-Blind (Evaluator) Primary Purpose: Treatment Duration: 12 weeks

ELIGIBILITY:
Inclusion Criteria

Experiencing hand arthralgia as a result of hormone therapy (aromatase inhibitors or tamoxifen) following breast cancer.

Ability to communicate pain levels effectively. Ability to follow simple instructions to participate in the intervention and assessments.

Exclusion Criteria Participants requiring any medication changes during the study period that could influence pain levels (increase or decrease).

Concurrent physiotherapy or occupational therapy specifically targeting the hand during the study.

Pre-existing diagnosis of arthritis or osteoarthritis in the hand before starting hormone therapy.

Presence of systemic diseases associated with hand arthralgia. Neurological conditions affecting hand movement.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | Pre Intervention and after the 8 weeks intervention
  A validated tool used to assess the severity of pain and its impact on daily functioning. Participants will report pain intensity on a numeric scale and describe how pain interferes with their daily life activities.

SECONDARY OUTCOMES:
DASH (Disabilities of the Arm, Shoulder, and Hand) Questionnaire | Pre Intervention and after the 8 weeks intervention
  A self-reported questionnaire that measures physical function and symptoms in individuals with upper limb conditions. It evaluates the ability to perform activities of daily living (ADLs) involving the hand, arm, and shoulder.
McCaffrey's Initial Pain Assessment Tool | Pre Intervention and after the 8 weeks intervention
  A structured assessment that includes diagrams for marking pain locations, along with descriptions of pain quality, intensity, and duration. It helps to capture a comprehensive view of pain perception.
ABILHAND Questionnaire | Pre Intervention and after the 8 weeks intervention
  A tool designed to assess manual ability and hand function in daily activities. Participants rate how easy or difficult it is to perform specific tasks requiring hand use.
Purdue Pegboard Test | Pre Intervention and after the 8 weeks intervention
  A standardized test to measure fine motor skills, hand-eye coordination, and manual dexterity. Participants are tasked with placing small pegs into holes on a board as quickly as possible, following a specified pattern.
Box and Block Test | Pre Intervention and after the 8 weeks intervention
  A test of gross manual dexterity where participants move small blocks from one compartment to another within a set time, assessing speed and motor function of the hand.
Minnesota Rate of Manipulation Test | Pre Intervention and after the 8 weeks intervention
  A comprehensive assessment of fine and gross manual dexterity, involving tasks like placing, rotating, and moving objects with one or both hands. It measures speed, accuracy, and coordination in manipulative tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Vanesa Abuín-Porras, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrod, Villaviciosa de Odón, Spain

IPD SHARING:
Plan to Share IPD: No